CLINICAL TRIAL: NCT04630977
Title: Long-term Intervention Effects of a Personalized, Home-based Exercise Program and Nutritional Advice, Along With the Inclusion of a Pre-workout Multi-ingredient Supplement on the Body Composition, Functional Capacity and Quality of Life of Middle-aged and Older Adults (40-70 Years)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Greenwich (Other)
Collaborators: Ingesport Health Spa Consulting (Unknown)
Responsible Party: Principal Investigator, Joel Puente, Principal Investigator, University of Greenwich
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UGreenwich2
Record Dates: First submitted 2020-11-08; First posted 2020-11-16 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Muscle Loss; Obesity; Obesity, Abdominal; Weight Loss; Happiness; Quality of Life; Self-Perception; Stress, Psychological
Keywords: Weight Loss; Body Composition; Home-Based; Supplement; Multi-ingredient
MeSH Terms: conditions — Muscular Atrophy; Obesity; Obesity, Abdominal; Weight Loss; Stress, Psychological | interventions — Nutritional Status; Diet, Healthy

STUDY DESIGN:
Intervention Model Description: One group will intake a pre-workout multi-ingredient supplement. The second group will intake an isocaloric placebo containing only carbohydrates.
  The third group (control) will take a non-caloric placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Every participant will be randomized to any of the groups. The principal investigator will be blinded for the supplement and allocation of the participants until the end of the analysis of the results after the intervention. Therefore, an external and third researcher will send the supplements to every participant and will keep the record of the randomised allocation of each of them until the end of the analysis of the last outcomes assessments collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multi-Ingredient Pre-workout Supplement (Experimental): This group of participants will intake a multi-ingredient supplement around ~15 minutes before every workout.
  The nutritional information of the supplement is: ~90 Kcal. for 25g of powder: carbohydrates -isomaltulose, fructose, maltodextrin- 15 g, essential amino-acids -Beta-alanine: 2.5g, L-arginine AKG: 2.5g, L-Leucine: 800mg, Taurine: 500mg, L-citrulline: 500mg- 6.8 g, Creatine monohydrate: 2.0g, Guarana Extract: 800mg, total caffeine: 160mg, and Magnesium: 112.5mg.
  They will also follow a previously designed progressive resistance training (3 times a week, around 1 hour a day, consisting of different exercises).
  Also, they will receive a specific guideline with simple tips to improve their nutritional patterns.
  The training sessions and the nutritional guideline will be the same for the three groups.
  Interventions: Dietary Supplement: Multi-ingredient Pre-workout supplement; Other: Progressive Resistance Training; Behavioral: Nutritional Patterns Guideline
- Isocaloric Placebo (Active Comparator): This group of participants will intake an isocaloric (only carbohydrates: Maltodextrin) supplement comparator, around ~15 minutes before every workout.
  The nutritional information of the supplement is: ~90 Kcal. for 23g of powder.
  They will also follow a previously designed progressive resistance training (3 times a week, around 1 hour a day, consisting of different exercises).
  Also, they will receive a specific guideline with simple tips to improve their nutritional patterns.
  The training sessions and the nutritional guideline will be the same for the three groups.
  Interventions: Other: Progressive Resistance Training; Behavioral: Nutritional Patterns Guideline
- Control (Sham Comparator): These participants will drink a non-caloric admixture with the same taste, texture and flavour.
  They will also follow a previously designed progressive resistance training (3 times a week, around 1 hour a day, consisting of different exercises).
  Also, they will receive a specific guideline with simple tips to improve their nutritional patterns.
  The training sessions and the nutritional guideline will be the same for the three groups.
  Interventions: Other: Progressive Resistance Training; Behavioral: Nutritional Patterns Guideline

INTERVENTIONS:
Dietary Supplement: Multi-ingredient Pre-workout supplement — Every important issue has been detailed before.
  Other Names: Preworkout
  Arms: Multi-Ingredient Pre-workout Supplement
Other: Progressive Resistance Training — The information about it has been detailed in advance.
  Other Names: PRT; RT
Behavioral: Nutritional Patterns Guideline — This intervention has also been described in advance.
  Other Names: Nutrition; Healthy Eating

SUMMARY:
The purpose of this study is to analyse the potential benefits of ingesting a commercially available pre-workout multi-ingredient supplement providing ~90 Kcal. for 25g of powder: carbohydrates -isomaltulose, fructose, maltodextrin- 15 g, essential amino-acids -Beta-alanine -L-arginine AKG, L-Leucine, Taurine, L-citrulline- 6.8 g, Creatine monohydrate: 2g, Guarana Extract: 800mg, total caffeine: 160mg, and Magnesium: 112.5mg) vs Placebo CHO intake on body composition, physical performance, Happiness Score (specially designed by our sponsor company, including different self-reported and validated tests on their short form) and every workout: Self-perceived energy feeling and adherence to the intervention.

DETAILED DESCRIPTION:
The methodology will follow a Home-based, online, double-blinded, randomised, long-term design. The participants recruited will be active, middle-aged and older healthy adults. The supplement intake will be a Pre-workout supplement intake or a placebo intake. The exercise training will be a Progressive Resistance Training, with sessions of ~1 hour (3 times/week). The intervention will last for a minimum of one year and the possibility to prolong it to another one (two years of intervention) if the adherence to the treatment was higher to the 75% of the participants (of, at least, 85% of the training sessions and supplementation intake).

The outcomes that will be assessed are: Body composition (fat mass and fat-free mass), physical performance (short test designed by Go Fit Lab: single-leg standing balance, upper-body strength - maximum number of push-ups repetitions in 15 seconds -, lower-body mechanical power - vertical jump -, agility/velocity - 30 seconds of static running at maximum velocity -, recovery assessment - 60 seconds monitoring of heart rate after the previous test -), Happiness Score (designed by Go Fit, including different self-reported validated tests, such as: Par-Q+, ACSM Cardiovascular Risk Factors Questionnaire, SF-12 for quality of life and self-perceived health status, PSS-4 Stress and mental health, Pittsburgh Sleeping Quality test, PREDIMED test: adherence to Mediterranean diet eating patterns, and the IPAQ short form), and for every workout: Self-perceived energy feeling (Questionnaire: Energy Level, Fatigue, Alertness and Focus for the Task), Rate of Perceived Exertion (OMNI RES Scale and Borg Scale) and adherence to regular physical exercise practise, healthy nutritional patterns, and supplement intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (no current injuries or illnesses which may interfere with the project).
* Recreationally active adults (a minimum of 3 and a maximum of 5 days of training sessions per week: combining resistance and endurance).

Exclusion Criteria:

* Participants younger than 40 or older than 70 years old.
* Participants with hard injuries, disabilities or pathologies.
* People taking medication or other supplements which may interfere with the multi-ingredient pre-workout or the training sessions.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-28 (Estimated)

PRIMARY OUTCOMES:
Fat Mass | Through study completion, an average of 1 year.
  Assessment of the total adipose tissue via Bioelectrical Impedance.
Fat-free Mass | Through study completion, an average of 1 year.
  Assessment of the total lean mass via Bioelectrical Impedance.
Health Perception questionnaire | 6 weeks.
  Short Form of 12 questions.
  Higher scores mean better outcomes (score from 0 to 100).
Pittsburgh Sleep Quality Index | 6 weeks.
  Short Form of 4 questions.
  Higher scores mean better outcomes (score from 1 to 5).
Stress Level and Mental Health | 6 weeks.
  Short Form of 4 questions.
  Higher scores mean worse outcomes (score from 1 to 5).
Adherence to a Mediterranean Diet (PREDIMED questionnaire) | 6 weeks.
  Short Form of 4 questions.
  Higher scores mean better outcomes (score from 1 to 5).
International Physical Activity Questionnaire | 6 weeks.
  7 questions.
  Higher scores mean better outcomes (score from 1 to 5).
Single-Leg balance | 6 Weeks
  Standing in one leg only, be capable of holding the position for 15 seconds. Performed with the dominant leg at first and the non-dominant leg afterwards.
  Score from 1 to 15 (higher scores mean better outcomes).
Upper-Body push strength | 6 Weeks
  Number of push-ups in 15 seconds.
  The score will be the number of Push-Ups performed (higher scores mean better outcomes).
Lower-body mechanical power | 6 Weeks
  Jump height with countermovement.
  The jump will be performed from a standing position, lateral to the wall and jumping to touch the wall as high as possible (with chalk in their finger-prints to mark the height they touched the wall).
  The score will be the height of the jump (higher scores mean better outcomes).
Recovery | 6 Weeks
  Static running in 1m2 square as fast as possible for 30 seconds and immediately after, Heart Rate will be monitored for 1 minute
  The score will be the difference from the Maximum Heart Rate minus the Heart Rate after 1 minute recovery (higher scores mean better outcomes).

SECONDARY OUTCOMES:
Adherence to the treatment (regular training, supplement intake and healthy eating) | 6 weeks
  The compliance with the training and supplementation protocols will be measured constantly, as well as the healthy eating patterns. Those participants who have spent 7 days or more in a row without training or taking the supplement, as well as a final accomplishment of the 85% will be discarded from the final analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Naclerio, Dr, Study Director — University of Greenwich
Locations (1):
- University of Greenwich, Avery Hill Campus, Sparrows Farm. Avery Hill, London., United Kingdom, SE9 2BT, London, Avery Hill, London., United Kingdom